CLINICAL TRIAL: NCT06653582
Title: Effect of Postural Reeducation Versus Pelvic Floor Muscle Training on Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Sally Mohamed Saeed, Principal Investigator, Misr University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005133
Record Dates: First submitted 2024-10-19; First posted 2024-10-22 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postural reeducation (Experimental): They will receive a program of postural reeducation with a home program for 12 weeks.
  Interventions: Other: Postural reeducation
- Pelvic floor exercises (Experimental): They will receive a program of pelvic floor exercises with a home program for 12 weeks.
  Interventions: Other: Pelvic floor exercises

INTERVENTIONS:
Other: Postural reeducation — The program will include postural awareness, stretching, McKenzie's method, and manual therapy for 12 weeks.
  Arms: Postural reeducation
Other: Pelvic floor exercises — The program will include pelvic floor exercises for 12 weeks. Three sets of 10 long contractions will be performed, each sustained for 6-8 seconds, three times a day. After each contraction, participants will be asked to rest for the same period. Two series of 10 fast contractions will be recommended, consisting of short, quick exercises of 1- to 2-second contractions, followed by long, sustained exercises lasting 5-10 seconds.
  Arms: Pelvic floor exercises

SUMMARY:
The purpose of the study is to evaluate the effects of postural reeducation compared to pelvic floor muscle training on urinary incontinence (UI) symptoms, the impact of UI, and quality of life (QoL) in women experiencing stress urinary incontinence (SUI)

DETAILED DESCRIPTION:
The study is designed as a randomized- controlled trial. It will be carried out on women suffering from stress urinary incontinence referred after urology consultations to the Physiotherapy Clinic in Soad Kafafy hospital.

UI, particularly SUI, affects up to 28% of the population and occurs during activities like coughing or sneezing due to inadequate urethral closure pressure. The pelvic floor muscles play a critical role in supporting pelvic organs and maintaining continence. Pelvic floor dysfunction is a significant contributor to SUI. Postural dysfunction can increase mechanical stress and lead to pelvic floor dysfunction. Postural re-education techniques aim to correct imbalances and improve pelvic floor muscle activity, potentially alleviating SUI symptoms by restoring muscle efficiency and enhancing continence.

ELIGIBILITY:
Inclusion Criteria:

* Fifty females with stress urinary incontinence.
* Age of 30-40 years.
* Body mass index (BMI) > 30 kg/m2

Exclusion Criteria:

* Genital prolapse grade 3 or 4 based on Pelvic Organ Prolapse Quantification Classification (POP-Q).
* Overactive bladder (OAB)
* Functional impairment (Barthel scale <85 points).
* Neurological or cognitive impairment (mini mental examination <24 points).
* Any other type of urinary incontinence.
* Pregnancy.
* History of spinal, hip, knee or foot surgery, pelvic and abdominal surgery (including cesarean section)
* Smoking, chronic cough, history of respiratory diseases, osteoporosis (self-reported).

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-01-25 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Urinary incontinence (UI) symptoms | 12 weeks
  UI symptoms will be measured using a 48-hour Pad Test [14]. This is a standardized test for assessing urine leakage that can be performed at home[15]. Women replace pads as needed over the course of 48 hours. The results are calculated by subtracting the net weight of used pads from the total weight of non-used pads. The Pad Test results can be classified as mild (4-20 g), moderate (21-74 g), or severe UI (> 75 g).
Urinary incontinence (UI) impact | 12 weeks
  It will be assessed using the International Consultation Incontinence Short-Form (ICIQ-UI-SF). UI impact will be derived from the values of the third question assessing overall impact ("How much does leaking urine interfere with everyday life?", ranging from 0 to 10), with a higher score indicating a greater UI impact.

SECONDARY OUTCOMES:
Urinary incontinence-Quality of life (UI-QoL) | 12 weeks
  It will be assessed using the International Consultation Incontinence Short-Form (ICIQ-UI-SF). The UI-QoL will be calculated using the questionnaire's final score (range from 0 to 21), which is the total of the three items, with a higher score indicating more severe UI and a bigger influence on QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Sally Mohamed Saeed, PhD, Principal Investigator — Lecturer, MUST university; Malak Adel Elmahdy, PhD, Principal Investigator — Lecturer, Al Hayah university
Locations (1):
- Faculty of physical therapy, MUST University, Giza, Egypt